CLINICAL TRIAL: NCT02216500
Title: Precision Ketogenic Therapy Effects on Electrical and Metabolic Abnormalities in Epilepsy
Brief Title: Ketogenic Therapy Effects on Electrical and Metabolic Abnormalities in Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201500942; OCR25124 (Other: UF OnCore)
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Seizures
Keywords: Ketogenic Therapy; Ketogenic Diet
MeSH Terms: conditions — Seizures | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Therapy (Experimental): Ketogenic Therapy will be administered.
  Interventions: Dietary Supplement: Ketogenic Therapy

INTERVENTIONS:
Dietary Supplement: Ketogenic Therapy — Ketogenic Therapy is based on a ratio of fat: protein+carbohydrate in which protein intake is adequate, fat intake is high, and carbohydrate intake is minimal.
  Other Names: Ketogenic Diet

SUMMARY:
Approximately a fourth of children with seizures do not respond adequately to available therapy. Ketogenic therapy has a long history as treatment for intractable epilepsy, but there is no agreement concerning how it works and what is the best way to administer it. This natural history study will collect data pertaining to both questions.

DETAILED DESCRIPTION:
The basis of Ketogenic Therapy is an altered macronutrient intake. It is based on a ratio of fat: protein+carbohydrate in which protein intake is adequate and carbohydrate is minimal. On Ketogenic Therapy, the body metabolizes fat, producing ketones as an energy source for the brain. Induction of ketosis has been shown to correlate with the reduction of seizures observed with Ketogenic Therapy. A major challenge of Ketogenic Therapy in children is that the compounds provided to stop seizure activity are the same compounds provided for growth and development. The altered macronutrient ratio that is the basis of Ketogenic Therapy is also a potential risk factor for dyslipidemia and may adversely affect growth. The investigators will evaluate efficacy of Ketogenic Therapy by assessing seizures and requirements for antiepileptic drugs. The investigators will evaluate adverse effects of Ketogenic Therapy by assessing dyslipidemia and growth. The investigators will foster optimal daily administration of therapy with structured training programs for caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose physician has prescribed the ketogenic diet
* Patients with lab tests consistent with the ability to metabolize a high fat and low carbohydrate diet
* Patients that can be compliant with administration of the therapy and with record keeping.

Exclusion Criteria:

* Patients with lab tests consistent with the inability to metabolize a high fat and low carbohydrate diet
* Patients at risk of being non-compliant with administration of the therapy and with record keeping

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2006-09; Primary Completion 2030-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Reduced seizures | 2 years
  Seizures will be charted from collected data.

SECONDARY OUTCOMES:
Reduced requirement for medications | 2 years
  Medication will be charted from collected data.

CONTACTS AND LOCATIONS:
Overall Officials: Peggy R. Borum, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States